CLINICAL TRIAL: NCT07254442
Title: Investigation of the Impact of Medications Used in COVID-19 Treatment and COVID-19 Vaccine on Hearing
Status: Completed | Type: Observational
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Azize Arzu KÖROĞLU KOÇYİĞİT, Audiologist, Lecturer, Zonguldak Bulent Ecevit University
Other Study IDs: 2021/61-18; 1919B012102481 (Other Grant/Funding Number: TUBİTAK)
Record Dates: First submitted 2025-09-26; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Hearing; COVID - 19; Ototoxicity
MeSH Terms: conditions — COVID-19; Ototoxicity | interventions — Hearing Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Control group: Group that has not had Covid-19
  Interventions: Diagnostic Test: Hearing tests
- Medication Group: The group that had Covid-19 and used medication
  Interventions: Diagnostic Test: Hearing tests
- Non-medication group: The group that had Covid-19 and did not use medication
  Interventions: Diagnostic Test: Hearing tests

INTERVENTIONS:
Diagnostic Test: Hearing tests — Participants' pure tone thresholds, high frequency thresholds, and otoacoustic emissions measurements were evaluated.

SUMMARY:
Investigation of the Impact of Medications Used in COVID-19 Treatment and COVID-19 Vaccine on Hearing

DETAILED DESCRIPTION:
This study aims to investigate the impact of medications containing the active ingredients hydroxychloroquine and favipiravir on the auditory system, as well as to examine the effect of COVID-19 on hearing and its potential relationship with medication use and COVID-19 vaccine dose.

ELIGIBILITY:
Inclusion Criteria:

Age between 18 and 35 For the Medication group: Having had COVID-19 and using COVID-19 medications For the Non-Medication group: Having had COVID-19 and not using COVID-19 medications For the Control group: Having never had COVID-19

Exclusion Criteria:

Previously diagnosed with hearing loss Use of ototoxic medications other than those specified Pathology detected during tympanometric evaluation or otoscopic examination Chronic disease Family history of hearing loss History of meningitis Neurological disorders Acute or chronic ear infection Admission to intensive care

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 1. Those who have had COVID-19 and are taking medication
  2. Those who have had COVID-19 and are not taking medication
  3. Healthy individuals who have not had COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Pure tone and high frequency hearing thresholds | December, 2021-February 2022
Transient evoked otoacoustic emissions - Signal/noise ratio | December, 2021-February 2022
Distortion product otoacoustic emissions- signal/noise ratio | December, 2021-February 2022

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No